CLINICAL TRIAL: NCT03370406
Title: Phase I, Dual Arm, Open-Label, Trial of Intralesional 5-Fluorouracil (5FU) and Intralesional 5FU Combined With Topical Calcipotriene in Patients With Squamous Cell Carcinoma (SCC) of the Lower Extremities
Brief Title: Intralesional 5-Fluorouracil (5FU), Topical Calcipotriene Treatment for SCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Melissa Pugliano-Mauro (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Melissa Pugliano-Mauro, Assistant Professor of Dermatology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19090229; 5P50CA121973-10 (NIH)
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Squamous Cell; Carcinoma; Lower Extremities; 5-Fluorouracil; Imiquimod
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — Fluorouracil; calcipotriene

STUDY DESIGN:
Intervention Model Description: 10 participants will serve as a control group, and will receive neither 5FU injection nor topical calcipotriene. 10 participants will receive one 1ml intralesional injection of 50mg/ml 5FU aqueous injectable solution once a month for 3 months. 10 participants will receive intralesional 5FU as in the previous group, additionally they will also apply 0.005% calcipotriene two (2) times daily for four (4) days one (1) day after each of three (3) 5FU injections to the same lesion. At the end of week eight (8), a 2mm punch biopsy of the lesion will be obtained for mid-point analysis, and will be stored for tissue banking. Four weeka after the last injection (week 12), the lesion will be surgical resected in all participants including the control group, to render the participants disease free. Resection is the current standard of care. A portion of the resected tumor and skin will also be stored for tissue banking, for future study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (No Intervention): Control group will receive neither 5-fluorouracil (5FU) injection nor topical 0.005% calcipotriene cream. This group will receive standard of care only. Lesion will be surgical resected on day 84 of study.
- 5FU Group (Experimental): 5-fluorouracil (5FU) Group participants will receive a 1ml intralesional injection of 5FU 50mg/ml aqueous injectable solution. One injection will be administered once monthly for 3 month. Injections will occur on d0, d28, and d56. Standard of care will be administered on d84 of study and lesion will be surgical resected.
  Interventions: Drug: 5-fluorouracil
- 5FU + 0.005% Calcipotriene cream Group (Experimental): 5-fluorouracil (5FU) + 0.005% calcipotriene cream Group participants will receive intralesional 5FU as in the previous group, additionally participants will also receive two (2) times daily for four (4) days one (1) day after each of three (3) 5FU injections topical application of 0.005% calcipotriene cream to the same lesion. Standard of care will be administered on d84 of study and lesion will be surgical resected.
  Interventions: Drug: 5-fluorouracil; Drug: Calcipotriene

INTERVENTIONS:
Drug: 5-fluorouracil — Intralesional injections of 50mg/ml over a 3 week period.
  Other Names: Adrucil; Tolak; Efudex; Carac; Fluoroplex; PremierPro Rx Fluorouracil; Fluorouracil Novaplus; 5FU
  Arms: 5FU + 0.005% Calcipotriene cream Group; 5FU Group
Drug: Calcipotriene — Topical application of .005% cream two (2) times daily for four (4) days one (1) day after each of three (3) 5FU injections..
  Other Names: Dovonex; Calcitrene; Sorilux; Calsodore; Kalosar
  Arms: 5FU + 0.005% Calcipotriene cream Group

SUMMARY:
This clinical trial proposes to evaluate a relatively unexplored approach to treatment of squamous cell carcinoma (SCC) on the lower extremities. The strategy is to directly and specifically deliver drug to the tumor. For the proposed phase I clinical trial, the investigators will perform intralesional injections of a well characterized, potent chemotherapeutic agent 5-fluorouracil (5FU) with and without a topical application of 0.005% calcipotriene cream to kill topically accessible SCC cells. The goal of the study is to evaluate the safety profile and tolerability of intralesional-5FU with and without a concomitant topical calcipotriene and measure the clinical objective response rate (ORR) in treated lesions compared to untreated lesions 3 weeks after treatment.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the skin is a common form of keratinocyte skin cancer. The majority of cutaneous SCCs occur on the head and neck, more so in men than women, but can occur anywhere squamous cells are found. Squamous cell carcinoma of the skin is usually not life-threatening, though it can be aggressive in some cases, and is normally treated with minor surgery.

Squamous cell carcinoma (SCC) of the lower extremity is a distinct subset of cutaneous squamous cell carcinomas which tend to occur multiply in elderly women. Histopathological studies of lower extremity SCCs reveals that they tend to be well differentiated and have low incidence of perineural and lymphovascular invasion and are also less prone to metastasis. Minor surgery has been the standard of care for this subset of SCC but leads to many complications such as poor wound healing and postoperative infections. Furthermore, a phenomenon called eruptive postoperative SCC can occur, in which cytokines released during wound healing triggering secondary tumor formation in genetically predisposed cells surrounding the original SCC. Given that lower extremity SCCs are less aggressive but more prone to surgical complications when excised, we believe they may be good candidates for localized non-surgical treatment.

5-fluorouracil (5FU) is a well-studied and characterized chemotherapeutic agent that has been used systemically, topically and intralesionally for a variety of malignancies and conditions including many dermatologic abnormalities.

It has been used on and off label topically for the treatment of actinic keratosis, SCC, superficial basal cell carcinoma, extra-mammary Paget's disease confined to the epidermis, Bowen's disease, porokeratosis, and genital warts. Intralesionally it has been used off label for the treatment of keloids, knuckle pads, warts, hypertrophic scars, basal cell carcinoma, and keratoanthoma.

Reports of its use intralesionally in invasive cutaneous SCC, other than in keratoacanthomas, are very limited. We are aware of 3 such reports in the literature. In the largest study to date, 6 weekly intralesional injections of 5FU-epinephrine gel were performed on 23 patients with cutaneous SCC on various body sites, 22 (96%) of whom demonstrated histologically confirmed tumor clearance. This study, however, used a proprietary gel formulation which is not widely available. There are two other case reports of successful treatment of SCC with 6-8 intralesional injections of 5FU at weekly intervals. The three published studies injected 0.6ml to 2.4ml of 5FU, per each weekly session, at concentrations of 30mg/ml to 50mg/ml.

Calcipotriene is a synthetic form of vitamin D. It is FDA approved for the treatment of psoriasis. Calcipotriene binds to vitamin D receptors on skin cells and helps regulate the growth and differentiation of skin cells. It inhibits keratinocyte proliferation (cell growth) and enhances keratinocyte differentiation. Recently it has been shown that calcipotriene acts as topical immune response modulator through induction of thymic stromal lymphoprotein (TSLP) expression. TSLP is an epithelium-derived cytokine and a regulator of allergic inflammation in the skin. It has been shown by Shadmehr Demehri et.al. that TSLP released by barrier-defective skin in mice blocks cancer development by recruiting T cells to mount robust antitumor immunity in the skin. The adaptive immune response mounted by TSLP against cancer can eliminate cancerous lesions in the skin and prevent new lesions from developing.

A recent clinical trial conducted by Demehri showed that participants treated with topical 5FU and topical and topical calcipotriene showed a significant reduction in the number of actinic keratosis (face, scalp, & upper extremities) vs topical 5FU and vaseline. Furthermore, the cohort treated with 5FU and topical and topical calcipotriene remained SCC-free for more than 1,500 days suggesting the induction of tissue-resident memory T (trm) cells.

The purpose of the study is to evaluate this relatively unexplored approach to the treatment of SCC on the lower extremities and establish a non-surgical therapy to improve outcomes, eliminate the need for surgery and mitigate the occurrence of infections and secondary tumor eruptions.

Topical 5FU is approved for the treatment of superficial basal cell carcinoma smaller than 2cm in diameter and not located on the feet, hands or feet but cannot penetrate deep enough into the skin to be an effective treatment for SCC. For the proposed phase I clinical trial, we propose to increase tumor accessibility by delivering 5FU directly and specifically to the tumor through intralesional injections to kill accessible localized SCC cells.

5FU is currently in clinical use with a well-established safety profile. It is anticipated that intralesional injections of 5FU will enable direct and specific delivery of chemotherapy to the tumor, thereby reducing the potential for systemic toxicity. Further, intralesional injections of-5FU enable tumoral delivery of locally effective concentrations of 5FU using doses that are orders of magnitude below those used currently for the intravenous (IV) treatment of multiple malignancies.

5FU alone may not be enough eliminate all the tumor cells so we also propose to treat a group of patients with intralesional 5FU and 0.005% calcipotriene topical cream. The goal is to develop a synergistic effect and establish an immune response to the 5FU induced apoptotic SCC cells in order to kill off any remaining SCC cells not undergoing apoptosis. Also 5FU alone may not be as effective of a treatment as the combination therapy in the prevention of secondary tumor recurrence. It is hoped that the combination therapy will induce a memory response and reduce the incidence of secondary tumors.

Participants will have at least 1 SCC lesion greater 1cm and less than 2 cm in largest diameter, on their lower extremities. The clinical diagnosis of SCC will be confirmed histologically by a deep shave biopsy of less than half of the lesion. The remainder of the lesion will be used for intralesional injections of 5FU or intralesional 5FU/topical calcipotriene according to the following schema:

In this study, a total of 30 patients will be randomly assigned into 3 groups. Randomization will be conducted using the UPCI randomizer, which is maintained by the Biostatistics Facility of UPCI (https://randomize.upci.pitt.edu/randomizer/home.seam). Group 1: 10 patients will serve as a control group, and will receive neither 5FU injection nor topical calcipotriene. Group 2: 10 patients, will receive a single intralesional injection of 50mg of 5FU in 1ml aqueous injectable solution once a month for 3 months. Group 3: 10 patients will receive intralesional 5FU as administered in the previous group. They will also apply a topical application of 0.005% calcipotriene cream to the same lesion two (2) times daily for four (4) days one (1) day after each of three (3) 5FU injections. At the time of initial consent, a 2 mm punch biopsy of the lesion will be obtained. Half of biopsy will be stored for tissue banking and future study, while the other half will be sent for histological confirmation of SCC. A second 2 mm punch biopsy will be taken at 2 months for mid-point analysis. This will be stored for tissue banking and future study. A month after the last injection (week 12), the lesion will be surgical resected in all patients including the control group, to render the patients disease free. Resection is the current standard of care for these tumors. A part of, or all of, the resected tumor and surrounding skin will be stored for tissue banking and future study.

All lesions will be photographed and treatment response will be evaluated 4 weeks after the first 5FU injection prior to excision.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed SCC more than 1.0 cm and less than 2.0 cm in diameter in the lower extremities, defined as the knees and below.
* Subjects must have an expected survival of greater than or equal to12 months.
* Subjects must not be on any other investigational device/drug treatment.
* Subjects must to be willing to adhere to the instructions of the Investigator and his research team and sign an Informed Consent Form prior to entry into the study.
* Patient is ≥ 18 years of age on day of signing informed consent.
* Patient must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Female patient of childbearing potential has a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.
* Female patients enrolled in the study, who are not free from menses for > 2 years, post hysterectomy/oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity throughout the study, starting with the first dose of study drug at visit 1 through 120 days after the last dose of study drug. Approved contraceptive methods include for example: intra-uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception. Male patients must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* Patients with any evidence of nodal (Nx) and/or metastatic disease including distant subcutaneous and/or lymph node metastases.
* Patients with primary non-cutaneous SCC - such as nasopharyngeal SCC.
* Patient with history of receiving organ transplantation.
* Patients with history of iatrogenic systemic immunosuppression.
* Patients with a history of skin or other disorder(s),that in the opinion of the investigator, requires topical application of steroids and/or other creams/ointments.
* Patients with evidence of active infection - active and/or untreated hepatitis B/C, HIV, etc - requiring systemic therapy.
* Patients with a known history of autoimmune disease.
* Patients with the following cardiac co-morbidities including:

  * Baseline known prolongation of QT/QTc interval (QTc interval >500 msec).
  * Heart failure either on clinical examination (manifestations include ascites, cardiomegaly, dyspnea, edema, gallop rhythm, hepatomegaly, oliguria, pleural effusion, pulmonary edema, tachycardia) or based on known decreased left ventricular ejection fraction (LV EF) <50%.
  * Patients who have had chemotherapy, radioactive or biological cancer therapy within four weeks prior to the first dose of study drug, or who has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the adverse effects (AEs) due to cancer therapeutics administered more than four weeks earlier. Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients currently participating or who have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study drug.
* Patients expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Patients with a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years.

  ° The time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
* Patients who have previously had a severe hypersensitivity reaction to 5-fluorouracil or imiquimod.
* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders.
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or are not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Patients who are, at the time of signing informed consent, regularly using illicit drugs or are recently (within the last year) abusing illicit substances (including alcohol).
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Determine number of subjects experiencing Dose Limiting Toxicity (DLT) higher than grade 2, as defined by CTCAE v. 4.0 | 84 days
  To assess Dose Limiting Toxicities (DLT) of intralesional-5FU and intralesional 5FU combined with topical imiquimod in subjects after 3 weeks of treatment.
  Dose Limiting Toxicities (DLT) are defined as:
  Higher-than grade 2 hematologic or non-hematologic toxicity that is definitely, probably, or possibly related to intralesional 5FU administration and/or topical imiquimod application. The NCI common terminology criteria for adverse events (CTCAE) version 4.0 will be used.
  Based on the results of the previous studies on treating SCCs with 5FU injection or topical imiquimod, significant toxicities are not expected. Adverse reactions were limited to local site reactions such as treatment site pain, induration, erythema, edema.
  If a patient has a DLT, doses will be delayed if any Grade >2 toxicities are not resolved to Grade 1 by the time of the next dose.

SECONDARY OUTCOMES:
Asses clinical objective response rate | 84 days
  Measure reduction in tumor burden to assess clinical objective response rate (ORR) in treated lesions. Response will be evaluated using modified Composite Assessment of Index Lesion Severity (CAILS) criteria by bi-dimensional measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Pugliano-Mauro, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- St. Margaret Hospital Dermatology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (learned intermediary) identified for this purpose.
  To achieve aims in the approved proposal.
  Proposals may be submitted up to 36 months following article publication. Proposals should be directed to puglianomauroma@upmc.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years through RedCap.
URL: https://www.ctsiredcap.pitt.edu/redcap/

REFERENCES:
- [Background] Rosenberg AR, Tabacchi M, Ngo KH, Wallendorf M, Rosman IS, Cornelius LA, Demehri S. Skin cancer precursor immunotherapy for squamous cell carcinoma prevention. JCI Insight. 2019 Mar 21;4(6):e125476. doi: 10.1172/jci.insight.125476. eCollection 2019 Mar 21. PMID 30895944
- [Background] Cunningham TJ, Tabacchi M, Eliane JP, Tuchayi SM, Manivasagam S, Mirzaalian H, Turkoz A, Kopan R, Schaffer A, Saavedra AP, Wallendorf M, Cornelius LA, Demehri S. Randomized trial of calcipotriol combined with 5-fluorouracil for skin cancer precursor immunotherapy. J Clin Invest. 2017 Jan 3;127(1):106-116. doi: 10.1172/JCI89820. Epub 2016 Nov 21. PMID 27869649
- [Background] Kim C, Ko CJ, Leffell DJ. Cutaneous squamous cell carcinomas of the lower extremity: a distinct subset of squamous cell carcinomas. J Am Acad Dermatol. 2014 Jan;70(1):70-4. doi: 10.1016/j.jaad.2013.09.026. Epub 2013 Nov 5. PMID 24210370
- [Background] Solus JF, Murphy GF, Kraft S. Cutaneous Squamous Cell Carcinomas of the Lower Extremities Show Distinct Clinical and Pathologic Features. Int J Surg Pathol. 2016 Feb;24(1):29-36. doi: 10.1177/1066896915599058. Epub 2015 Aug 10. PMID 26261102
- [Background] Munday WR, Leffell DJ, McNiff JM, Ko CJ. Histopathologic features of multiple cutaneous squamous cell carcinomas of the lower extremity. J Cutan Pathol. 2016 Sep;43(9):759-65. doi: 10.1111/cup.12738. Epub 2016 Jun 14. PMID 27220356
- [Background] Bangash SJ, Green WH, Dolson DJ, Cognetta AB Jr. Eruptive postoperative squamous cell carcinomas exhibiting a pathergy-like reaction around surgical wound sites. J Am Acad Dermatol. 2009 Nov;61(5):892-7. doi: 10.1016/j.jaad.2009.01.037. Epub 2009 Sep 18. PMID 19766351
- [Background] Moore AY. Clinical applications for topical 5-fluorouracil in the treatment of dermatological disorders. J Dermatolog Treat. 2009;20(6):328-35. doi: 10.3109/09546630902789326. PMID 19954388
- [Background] Metterle L, Nelson C, Patel N. Intralesional 5-fluorouracil (FU) as a treatment for nonmelanoma skin cancer (NMSC): A review. J Am Acad Dermatol. 2016 Mar;74(3):552-7. doi: 10.1016/j.jaad.2015.09.040. Epub 2015 Nov 11. PMID 26577512
- [Background] Kraus S, Miller BH, Swinehart JM, Shavin JS, Georgouras KE, Jenner DA, Griffin E, Korey A, Orenberg EK. Intratumoral chemotherapy with fluorouracil/epinephrine injectable gel: a nonsurgical treatment of cutaneous squamous cell carcinoma. J Am Acad Dermatol. 1998 Mar;38(3):438-42. doi: 10.1016/s0190-9622(98)70502-x. PMID 9520026
- [Background] Reisinger DM, Cognetta AB Jr, Pynes LT, Paredes AA Jr, Sweeney TJ, Dolson DJ. Treatment of a giant squamous cell carcinoma on the dominant thumb with intralesional 5-fluorouracil. J Am Acad Dermatol. 2011 Jul;65(1):219-21. doi: 10.1016/j.jaad.2009.11.017. No abstract available. PMID 21679825
- [Background] Morse LG, Kendrick C, Hooper D, Ward H, Parry E. Treatment of squamous cell carcinoma with intralesional 5-Fluorouracil. Dermatol Surg. 2003 Nov;29(11):1150-3; discussion 1153. doi: 10.1046/j.1524-4725.2003.29355.x. PMID 14641346
- [Background] Love WE, Bernhard JD, Bordeaux JS. Topical imiquimod or fluorouracil therapy for basal and squamous cell carcinoma: a systematic review. Arch Dermatol. 2009 Dec;145(12):1431-8. doi: 10.1001/archdermatol.2009.291. PMID 20026854
- [Background] Peris K, Micantonio T, Fargnoli MC, Lozzi GP, Chimenti S. Imiquimod 5% cream in the treatment of Bowen's disease and invasive squamous cell carcinoma. J Am Acad Dermatol. 2006 Aug;55(2):324-7. doi: 10.1016/j.jaad.2006.04.004. PMID 16844522

DOCUMENTS (1):
  • Informed Consent Form (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03370406/ICF_003.pdf